CLINICAL TRIAL: NCT01348620
Title: Single Port Laparoscopic Cholecystectomy Versus Four Port Laparoscopic Cholecystectomy: Impact on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Dr Perantoni Laura, Sacro Cuore Don Calabria General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNT-2011
Record Dates: First submitted 2011-04-26; First posted 2011-05-05 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Postoperative Pain
Keywords: single port cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single port laparoscopic device (Experimental)
  Interventions: Device: Single port laparoscopic cholecystectomy SINGLE SITE LAPAROSCOPY ACCESS SYSTEM (Johnson & Johnson Medical Spa)
- Four-port laparoscopic device (Active Comparator)
  Interventions: Procedure: Four port laparoscopic cholecystectomy surgery

INTERVENTIONS:
Device: Single port laparoscopic cholecystectomy SINGLE SITE LAPAROSCOPY ACCESS SYSTEM (Johnson & Johnson Medical Spa) — Single port laparoscopic cholecystectomy. SINGLE SITE LAPAROSCOPY ACCESS SYSTEM (Johnson & Johnson Medical Spa)
  Other Names: One-trocar cholecistectomy
  Arms: Single port laparoscopic device
Procedure: Four port laparoscopic cholecystectomy surgery — Four port laparoscopic cholecystectomy surgery
  Other Names: traditional Laparoscopic cholecistectomy
  Arms: Four-port laparoscopic device

SUMMARY:
This is a single-institution, prospective, randomized controlled trial. Subjects determined to need a cholecystectomy will be consented for surgery and study participation prior to enrollment in this study. Patients will then be randomized to receive either a single port laparoscopic cholecystectomy or a four port laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The main advantages of laparoscopic surgery are reduced postoperative pain, shorter hospital stay and the cosmetic result. Although reduced, however, pain is still substantial and constitutes the main clinical problem after laparoscopic cholecystectomy, in particular for future daily planned procedures.

Recently, a new technique of laparoscopic cholecystectomy has been developed, in which all instruments are inserted through the same port placed in the umbilical incision. This technique for cholecystectomy has been proved to be feasible and safe by several studies.

The purpose of the study is to compare postoperative pain, operating time, cosmetic result, between one port and standard laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Biliary cholic
* Biliary dyskinesia
* Gallbladder polyps
* Other diagnosis at the discretion of the surgeon

Exclusion Criteria:

* History of Acute cholecystitis
* Jaundice
* Choledocolithiasis
* History of Pancreatitis
* Severe comorbidity
* BMI > 30

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain scores (visual analogue pain scale from 0-10) | Before surgery (baseline) and 2 hrs, 4 hrs, 6hrs, 12hrs, 24hrs and 48hrs after surgery

SECONDARY OUTCOMES:
Patient-assessed cosmesis on the Visual Analogue Scale | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sacro Cuore - Don Calabria Hospital, Negrar, Verona, Italy

REFERENCES:
- [Background] Rao PP, Bhagwat SM, Rane A, Rao PP. The feasibility of single port laparoscopic cholecystectomy: a pilot study of 20 cases. HPB (Oxford). 2008;10(5):336-40. doi: 10.1080/13651820802276622. PMID 18982149
- [Background] Hirano Y, Watanabe T, Uchida T, Yoshida S, Tawaraya K, Kato H, Hosokawa O. Single-incision laparoscopic cholecystectomy: single institution experience and literature review. World J Gastroenterol. 2010 Jan 14;16(2):270-4. doi: 10.3748/wjg.v16.i2.270. PMID 20066749
- [Background] Tacchino R, Greco F, Matera D. Single-incision laparoscopic cholecystectomy: surgery without a visible scar. Surg Endosc. 2009 Apr;23(4):896-9. doi: 10.1007/s00464-008-0147-y. Epub 2008 Sep 25. PMID 18815836
- [Background] Gumbs AA, Milone L, Sinha P, Bessler M. Totally transumbilical laparoscopic cholecystectomy. J Gastrointest Surg. 2009 Mar;13(3):533-4. doi: 10.1007/s11605-008-0614-8. PMID 18709515
- [Background] Kuon Lee S, You YK, Park JH, Kim HJ, Lee KK, Kim DG. Single-port transumbilical laparoscopic cholecystectomy: a preliminary study in 37 patients with gallbladder disease. J Laparoendosc Adv Surg Tech A. 2009 Aug;19(4):495-9. doi: 10.1089/lap.2008.0424. PMID 19630589
- [Derived] Partelli S, Barugola G, Sartori A, Crippa S, Falconi M, Ruffo G. Single-incision laparoscopic cholecystectomy versus traditional laparoscopic cholecystectomy performed by a single surgeon: findings of a randomized trial. Surg Today. 2016 Mar;46(3):313-8. doi: 10.1007/s00595-015-1182-7. Epub 2015 Jun 3. PMID 26036221
- [Derived] Steinemann DC, Raptis DA, Lurje G, Oberkofler CE, Wyss R, Zehnder A, Lesurtel M, Vonlanthen R, Clavien PA, Breitenstein S. Cosmesis and body image after single-port laparoscopic or conventional laparoscopic cholecystectomy: a multicenter double blinded randomised controlled trial (SPOCC-trial). BMC Surg. 2011 Sep 12;11:24. doi: 10.1186/1471-2482-11-24. PMID 21910897